CLINICAL TRIAL: NCT05250284
Title: The Intersection of Oncology Care and Worker Well-Being
Status: Recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute for Occupational Safety and Health (NIOSH/CDC) (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 21-4139.cc; U19OH011227 (NIH)
Record Dates: First submitted 2022-01-20; First posted 2022-02-22 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Solid Tumor
Keywords: Newly Diagnosed Primary Solid Tumor; Men; Employed; Chemotherapy; Oral Agent; Radiation Therapy
MeSH Terms: conditions — Multiple Endocrine Neoplasia Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: WellBQ — National Institue for Occupational Safety and Health Worker Well-Being Questionnaire is comprised of 21 scales (multiple items assessing a single construct) and 31 single items that cover worker well-being. Domains include (i) work evaluation and experience, (ii) workplace policies and culture, (iii) workplace physical environment and safety climate, (iv) health status, and (v) home, community, and society.
Behavioral: PROMIS — Patient-Reported Outcomes Measurement Information System is a set of person-centered measures that evaluates and monitors physical, mental, and social health in adults and children.

SUMMARY:
The goals of this study will be a greater understanding of cancer patients' well-being experience through the care/treatment continuum. An important aspect of the study is an understanding of work- and treatment-related challenges experienced by low-income men, many of whom will be Latino. At the 12-month observation period, the investigators will learn whether these men work long-term and how work status relates to well-being.

DETAILED DESCRIPTION:
Labor supply and well-being outcomes will be evaluated at 3 timepoints (baseline, start of treatment, 12 months). The likelihood of remaining employed will be estimated with linear probability models as is the convention in labor economics. The study team also estimate employment using analogous logistic models, reporting marginal effects. Weekly hours worked will be estimated using ordinary least squares regression. In addition to measuring raw hours, the team estimate change and percent change in hours worked from baseline. These models can be expanded to accommodate control variables for worksite and job characteristics as well as accommodations, satisfaction, and other covariates predictive employment and hours worked.

Well-being will be assessed as specified by the Worker Well-Being Questionnaire (WellBQ) Manual23 and Patient Reported Outcomes Measurement Information Systems (PROMIS) domains. For PROMIS, subjects respond to a 4-item questionnaire for each domain. Responses are summed and standardized to t-scores, with higher t-scores representing higher levels of the domain measured. For example, an individual with a PROMIS depression t-score of 50 is the average observed in the general U.S. population, while a t-score of 60 indicates one standard deviation above the average score in the general population and represents moderate depressive symptoms. Guided by previous health literature, the team consider a half standard deviation (5-point) increase from initial scores a meaningful improvement for all PROMIS domains. The literature also suggests that meaningful change ranges from 2 to 6 points. Secondary to Aim 1, the team will assess the correlation between PROMIS measures and WellBQ. The WellBQ is at an earlier stage of adoption, warranting side-by-side comparison with established instruments like PROMIS. The InCharge instrument will be evaluated as suggested by the developers.

ELIGIBILITY:
Inclusion Criteria:

* Males
* Ages 21 to 70
* Newly diagnosed with a first primary solid tumor
* colorectal, lung, and head and neck
* Currently employed (defined as working 10+ hours per week) with the intention to continue working or return to work
* Within 2 months of initiating infusion chemotherapy, oral agent, or radiation therapy

Ages: 21 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Study Population: sample consists of employed men newly diagnosed with a first primary solid tumor. define employed as working 10+ hours per week at diagnosis with the intention to continue working or return to work. Patients must be aged 21 to 70 years and within 2 months of initiating infusion chemotherapy, oral agent, or radiation therapy.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-04-04 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Employment Hours Worked | 2 years
  Employment and weekly hours worked will be assessed using questions from the Current Population Survey (CPS)
Worker Well-being | 2 years
  Worker well-being will be measured by the NIOSH WellBQ
Psychosocial Outcomes of Employed Males with Cancer using the validated Stress Thermometer. | 2 years
  Depression and anxiety will be measured using the well-validated Stress Thermometer, a single item tool using a 0 (no distress) to 10 (extreme distress) - point Likert scale resembling a thermometer.
Psychosocial Outcomes of Employed Males with Cancer using PROMIS domains | 2 years
  Psychosocial outcomes will be measured using the validated PROMIS domains. Subjects respond to a 4-item questionnaire for each domain. Responses are summed and standardized to t-scores, with higher t-scores representing higher levels of the domain measured. For example, an individual with a PROMIS depression t-score of 50 is the average observed in the general U.S. population, while a t-score of 60 indicates one standard deviation above the average score in the general population and represents moderate depressive symptoms.
Financial Burden of Employed Males with Cancer | 2 yearas
  A systematic review of methods for measuring financial burden following cancer treatment identified 6 subdomains that represent perceptions of and reactions to financial distress: (i) financial spending, (ii) use of passive financial resources, (iii) psychosocial responses, (iv) support seeking, (v) coping with care or (vi) coping with ones' lifestyle.64 We chose the InCharge Financial Well-being/Financial Distress Scale (8 items) that covers most domains and is widely used in cancer patients.

CONTACTS AND LOCATIONS:
Overall Officials: Cathy Bradley, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided